CLINICAL TRIAL: NCT00550550
Title: A Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study Evaluating the Efficacy and Safety of Sublingual Immunotherapy With SCH 697243 (Phleum Pratense) in Children 5 to <18 Years of Age With a History of Grass Pollen Induced Rhinoconjunctivitis With or Without Asthma
Brief Title: Efficacy and Safety of Grass Sublingual Tablet in Children and Adolescents (P05239 AM3)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05239; 3733251
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Results first posted 2012-09-07 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Rhinoconjunctivitis; Rhinitis; Conjunctivitis; Allergy
Keywords: rhinoconjunctivitis; rhinitis; conjunctivitis; allergy; allergen; immunotherapy
MeSH Terms: conditions — Rhinitis; Conjunctivitis; Hypersensitivity | interventions — Loratadine; Olopatadine Hydrochloride; Mometasone Furoate; Albuterol; Fluticasone; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo; Drug: Loratadine Syrup 1 mg/mL Rescue Treatment; Drug: Loratadine 10 mg Rescue Treatment; Drug: Olopatadine 0.1% Rescue Treatment; Drug: Mometasone furoate 50 mcg Rescue Treatment; Drug: Albuterol 108 mcg Rescue Treatment; Drug: Fluticasone 44 mcg Rescue Treatment; Drug: Prednisone 5 mg Rescue Treatment
- SCH 697243 (Experimental): Grass Sublingual Tablet (Phleum pratense extract)
  Interventions: Biological: SCH 697243; Drug: Loratadine Syrup 1 mg/mL Rescue Treatment; Drug: Loratadine 10 mg Rescue Treatment; Drug: Olopatadine 0.1% Rescue Treatment; Drug: Mometasone furoate 50 mcg Rescue Treatment; Drug: Albuterol 108 mcg Rescue Treatment; Drug: Fluticasone 44 mcg Rescue Treatment; Drug: Prednisone 5 mg Rescue Treatment

INTERVENTIONS:
Drug: Placebo — Placebo sublingual tablet, once daily
  Arms: Placebo
Biological: SCH 697243 — Grass sublingual tablet, once daily
  Other Names: Phleum pratense extract
  Arms: SCH 697243
Drug: Loratadine Syrup 1 mg/mL Rescue Treatment — Loratadine Syrup 1 mg/mL was dosed orally once daily at a dose of 5 mg for children aged 5 to <6 years of age and at a dose of 10 mg for children aged 6 to <18 years of age as rescue medication for symptoms of rhinoconjunctivitis among participants with a total symptom score ≥4.
  Other Names: Claritin
Drug: Loratadine 10 mg Rescue Treatment — Loratadine 10 mg RediTabs tablets were dosed orally once daily at a dose of 10 mg for children aged 6 to <18 years of age as rescue medication for symptoms of rhinoconjunctivitis among participants with a total symptom score ≥4.
  Other Names: Claritin
Drug: Olopatadine 0.1% Rescue Treatment — Olopatadine hydrochloride 0.1% ophthalmic solution was dosed intraocularly at a dose of 1 drop in each affected eye twice daily, in addition to loratadine, as rescue medication for participants with persistent eye symptoms due to rhinoconjunctivitis.
  Other Names: Pantanol
Drug: Mometasone furoate 50 mcg Rescue Treatment — Mometasone furoate monohydrate nasal spray 50 mcg was dosed intranasally at a dose of one spray in each nostril once daily for participants aged 5 to <12 years and a dose of 2 sprays in each nostril once daily for participants aged 12 to <18 years as rescue medication for nasal symptoms of rhinoconjunctivitis among participants with a total symptom score of ≥4 despite loratadine and mometasone furoate nasal spray.
  Other Names: Nasonex
Drug: Albuterol 108 mcg Rescue Treatment — Albuterol sulfate inhalation aerosol 108 mcg/inhalation was administered via inhalation at a dose of 2 inhalations every 4 to 6 hours as rescue medication among participants aged 5 to <18 years with asthma symptoms .
  Other Names: Proventil; Ventolin; Volmax; Vospire
Drug: Fluticasone 44 mcg Rescue Treatment — Fluticasone propionate inhalation aerosol 44 mcg/inhalation was administered via inhalation at a dose of 2 inhalations twice daily among participants aged 12 to <18 years up to a maximum dose of 10 inhalations twice daily, in combination with albuterol, among participants with ≥4 albuterol sulfate inhalations/day for 2 days as rescue medication for nocturnal asthma or shortness of breath.
  Other Names: Flonase
Drug: Prednisone 5 mg Rescue Treatment — Prednisone tablet 5 mg was administered orally at a dose of 1 mg/kg/day once daily up to a maximum of 50 mg/day on Day 1, and at a dose of 0.5 mg/kg/day once daily up to a maximum of 25 mg/day on Days 2, 3, 5, and 7 as rescue medication for asthma exacerbation at the discretion of the investigator.
  Other Names: Deltasone; Meticorten; Orasone; Prednicen-M; Prednicot; Sterapred; Sterapred DS

SUMMARY:
The purpose of the study is to investigate the efficacy and safety of a grass sublingual tablet in children and adolescents with a history of grass-pollen induced rhinoconjunctivitis with or without asthma.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group study in participants aged 5 to <18 years of either sex, and of any race with a history of grass pollen induced rhinoconjunctivitis with or without asthma. While receiving treatment, participants will receive either grass sublingual tablet or placebo. Open-label rescue medications for the rhinoconjunctivitis and asthma symptoms will be provided. Participants will visit the study site for at least 12 visits. A total of 10 allergic symptoms, 6 rhinoconjunctivitis and 4 lung symptoms, will be recorded daily on an electronic diary by the participant/parent/guardian.

The start and end of the grass pollen season (GPS) was determined based on the regional grass pollen count, and lasted up to 162 days. For each region, the GPS is defined as the first day of 3 consecutive recorded days with a grass pollen count of ≥ 10 grains/m^3, to the last day of the last occurrence of 3 consecutive recorded days with a grass pollen count ≥ 10 grains/m^3, inclusively.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 5 to <18 years of age, of either sex, and of any race.
* Participant must have a clinical history of significant allergic rhinoconjunctivitis to grass (with or without asthma) diagnosed by a physician and have received treatment for their disease during the previous GPS.
* Participant must have a positive skin prick test response (average wheal diameter >=5 mm larger than the saline control after 15 to 20 minutes) to Phleum pratense at the Screening Visit.
* Participant must have positive specific IgE against Phleum pratense (>= IgE Class 2) at the Screening Visit.
* Participant must have an FEV1 >=70% of predicted value at the Screening Visit.
* A participant's safety laboratory tests and vital signs conducted at the Screening Visit must be within normal limits or clinically acceptable to the investigator/sponsor.
* A participant (and/or parent/guardian for subjects under the age of legal consent or who otherwise are unable to provide independent consent) must be willing to give written informed consent/assent and be able to adhere to dose and visit schedules.
* Female participants of childbearing potential must be using a medically acceptable and adequate form of birth control. These include:

  * hormonal contraceptives as prescribed by a physician (oral, hormonal vaginal ring, hormonal implant or depot injectable);
  * medically prescribed intra-uterine device;
  * medically prescribed topically-applied transdermal contraceptive patch;
  * double-barrier method (eg, condom in combination with a spermicide); vasectomy and tubal ligation should each be considered as single barrier.
* Female participants of childbearing potential should be counseled in the appropriate use of birth control while in the study. Female participants who are not currently sexually active must agree and consent to use one of the above-mentioned methods if they become sexually active while participating in the study.
* Female participants of childbearing potential must have a negative urine pregnancy test at the Screening Visit in order to be considered eligible for enrollment.

Exclusion Criteria:

* Participant with a clinical history of symptomatic seasonal allergic rhinitis and/or asthma, having received regular medications due to another allergen during or potentially overlapping the GPS.
* Participant with a clinical history of significant symptomatic perennial allergic rhinitis and/or asthma having received regular medication due to an allergen to which the participant is regularly exposed.
* Participant with sufficient pre-seasonal data in the observational phase will not be eligible to continue in the treatment phase if the participant: 1) does not experience an increase in rhinoconjunctivitis symptom score of equal to or greater than 4 above the pre-seasonal average symptom score for at least 2 days, 2) does not use allergy rescue medication for at least 2 days, during the observational phase Year 1 2008 GPS.
* Participant has received an immunosuppressive treatment within 3 months prior to the Screening Visit (except steroids for allergic and asthma symptoms).
* Participant with a clinical history of severe asthma.
* Participant with history of anaphylaxis with cardiorespiratory symptoms.
* Participant with history of self-injectable epinephrine use.
* Participant with a history of chronic urticaria and angioedema.
* Participant with clinical history of chronic sinusitis during the 2 years prior to the Screening Visit.
* Participant with current severe atopic dermatitis.
* Female participants who are breast-feeding, pregnant, or intending to become pregnant.
* Participant who has had previous treatment by immunotherapy with grass pollen allergen or any other allergen within the 5 years prior to the Screening Visit.
* Participant with a known history of allergy, hypersensitivity or intolerance to the ingredients of the IMP (except for Phleum pratense), rescue medications, or self-injectable epinephrine.
* Participant with any clinically significant condition or situation, other than the condition being studied that, in the opinion of the investigator, would interfere with the study evaluations or optimal participation in the study. Specific examples include but are not limited to hypertension being treated with beta blockers, coronary artery disease, arrhythmia, stroke, ocular conditions requiring topical beta blockers, any condition requiring the use of beta blockers.
* Participant who has used any investigational drugs within 30 days of the Screening Visit.
* Participant who is participating in any other clinical study.
* Participant who is a family member of the investigational study staff conducting this study.
* Participant who is unable to meet medication washout requirements as listed in the protocol.
* Participant who is unlikely to be able to complete the trial, for any reason, or likely to travel for extended periods of time during the GPS, which in the opinion of the investigator will compromise the data.
* Participant with a clinically significant abnormal vital sign or laboratory value that would preclude participation in the study.
* A participant participating in this study may not participate in this same study at another investigational site.
* A participant must not be randomized into this study more than once.
* Participant who is unable to or will not comply with the use of self-injectable epinephrine.
* Participants who may be at greater risk of developing adverse reactions after epinephrine administration.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 345 (Actual)
Dates: Start 2007-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

REFERENCES:
- [Result] Blaiss M, Maloney J, Nolte H, Gawchik S, Yao R, Skoner DP. Efficacy and safety of timothy grass allergy immunotherapy tablets in North American children and adolescents. J Allergy Clin Immunol. 2011 Jan;127(1):64-71, 71.e1-4. doi: 10.1016/j.jaci.2010.11.034. PMID 21211642
- [Derived] Hebert J, Blaiss M, Waserman S, Kim H, Creticos P, Maloney J, Kaur A, Li Z, Nelson H, Nolte H. The efficacy and safety of the Timothy grass allergy sublingual immunotherapy tablet in Canadian adults and children. Allergy Asthma Clin Immunol. 2014 Oct 30;10(1):53. doi: 10.1186/1710-1492-10-53. eCollection 2014. PMID 25685162

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 345 subjects were randomized at a total of 68 sites (58 sites from United States; 10 sites from Canada) to treatment assignment, and 344 subjects received at least one dose of study medication.
Groups:
- SCH 697243: SCH 697243 (Phleum pratense extract) administered sublingually once daily.
- Placebo: Matching placebo tablet administered sublingually once daily.
Period: Overall Study
Arm/Group | SCH 697243 | Placebo
Started | 176 | 169
Number Treated | 175 | 169
Completed | 142 | 140
Not Completed | 34 | 29
Not completed — Adverse Event | 13 | 5
Not completed — Treatment Failure | 0 | 1
Not completed — Lost to Follow-up | 4 | 0
Not completed — Withdrawal by Subject | 10 | 8
Not completed — Protocol Violation | 5 | 14
Not completed — Did Not Meet Protocol Eligibility | 1 | 1
Not completed — Randomized But Not Treated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SCH 697243 | Placebo | Total
Number analyzed (Participants) | 175 | 169 | 344
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.1 (3.0) | 12.6 (3.0) | 12.3 (3.0)
Gender [Count of Participants; unit: Participants]
  Female | 57 | 64 | 121
  Male | 118 | 105 | 223

OUTCOME MEASURES:

1. Primary Outcome: Participant Total Combined Symptom (TCS) Score Over the Entire Grass Pollen Season (GPS)
Description: The TCS is the sum of the rhinoconjunctivitis daily symptom score (DSS) and rhinoconjunctivitis daily medication score (DMS) averaged over the entire GPS. The TCS ranged from 0 (no symptoms and no rescue medication use) to 54 (most severe symptoms and maximum use of rescue medication), with increasing score indicating a higher level of symptom severity. The DSS is composed of 6 rhinoconjunctivitis symptoms with scores from 0 (best) to 18 (worst), with increasing score indicating increased severity. The DMS is composed of a sum of the scores associated with rescue medication use per day. The range for the DMS was 0 (no rescue medication use) to 36 (maximum use of rescue medication), with a lower score indicating less use of rescue medication.
Time Frame: From the Start of the GPS to the End of the GPS
Population: The Full Analysis Set (FAS) population was comprised of all participants randomized with at least one post-treatment diary data entry.
Measure: Mean (Standard Error); unit: Units on a Scale
Groups:
- SCH 697243: Rapidly dissolving grass pollen allergen tablet administered sublingually once daily.
- Placebo: Rapidly dissolving matching placebo tablet administered sublingually once daily.
Arm/Group | SCH 697243 | Placebo
Number analyzed (Participants) | 149 | 158
Units on a Scale | 4.62 (0.52) | 6.25 (0.51)
Statistical Analysis 1: Comparison: SCH 697243 vs Placebo; Test type: Superiority or Other; p = 0.001, ANOVA; Asthma status, treatment group, and site were fixed effects; Mean Difference (Final Values) = -1.63, 95% CI 2-sided [-2.60 to -0.66]

2. Secondary Outcome: Participant Average Rhinoconjunctivitis Daily Symptom Scores (DSS) Over the Entire GPS
Description: The DSS is composed of six rhinoconjunctivitis symptoms which were recorded daily including runny nose, blocked nose, sneezing, itchy nose, gritty feeling/red/itchy, and watery eyes, and the symptoms were measured on a scale of 0 (no symptom) to 3 (severe symptoms). A higher score indicated a higher level of symptoms and the total daily score could range from 0 (best) to 18 (worst).
Time Frame: Start of the GPS to the End of the GPS
Population: The FAS population was comprised of all participants with at least one post-treatment diary data entry.
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | SCH 697243 | Placebo
Number analyzed (Participants) | 149 | 158
Units on a Scale | 3.71 (0.40) | 4.91 (0.41)
Statistical Analysis 1: Comparison: SCH 697243 vs Placebo; Test type: Superiority or Other; p = 0.005, ANOVA; Asthma status, treatment group, and site were fixed effects; Mean Difference (Final Values) = -1.20, 95% CI 2-sided [-1.95 to -0.45]

3. Secondary Outcome: Participant Average Rhinoconjunctivitis Daily Medication Score (DMS) Over the Entire GPS
Description: The DMS is composed of a sum of the scores associated with rescue medication use per day. Rescue medications were implemented when a participant had a symptom score >= 4. Rescue medications for allergic rhinoconjunctivitis were to be utilized in a step-wise fashion: loratadine, olopatadine hydrochloride 0.1% opthalmic solution, mometasone, and prednisone, in that sequence. The score for the DMS ranged from 0 (no use of rescue medication) to 36 (maximum use of rescue medication). A lower medication score indicated less impact on symptoms and was suggestive of less use of rescue medication.
Time Frame: Start of the GPS to the End of the GPS
Population: The FAS population was comprised of all participants randomized with at least one post-treatment diary data entry.
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | SCH 697243 | Placebo
Number analyzed (Participants) | 149 | 158
Units on a Scale | 0.91 (0.25) | 1.33 (0.23)
Statistical Analysis 1: Comparison: SCH 697243 vs Placebo; Test type: Superiority or Other; p = 0.066, ANOVA; Asthma status, treatment group, and site were fixed effects; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.88 to 0.03]

4. Secondary Outcome: Participant Average Weekly Rhinoconjunctivitis Quality-of-Life Questionnaire (RQLQ) Total Score Over the Entire GPS
Description: The RQLQ has 28 questions and focusses on 7 domains that may be significantly impaired in participants with seasonal allergic rhinoconjunctivitis: sleep impairment, non-nasal symptoms, practical problems, nasal symptoms, eye symptoms, activity limitations, and emotional difficulty. The RQLQ score is the mean of all 28 responses and the individual domain scores are the means of the items in those domains. RQLQ scores range from 0 (best) to 6 (worst), with a higher score indicating more significant impairment.
Time Frame: Start of the GPS to the End of the GPS
Population: The FAS population was comprised of all participants randomized with at least one post-treatment diary data entry for the rhinoconjunctivitis quality-of-life measure.
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | SCH 697243 | Placebo
Number analyzed (Participants) | 109 | 111
Units on a Scale | 1.45 (0.11) | 1.77 (0.12)
Statistical Analysis 1: Comparison: SCH 697243 vs Placebo; Test type: Superiority or Other; p = 0.042, ANOVA; Asthma status, treatment group, and site were fixed effects; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-0.60 to -0.03]

ADVERSE EVENTS:
Arm/Group | SCH 697243 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/176 | 4/169
Other Adverse Events (participants affected / at risk) | 141/176 | 121/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCH 697243 (N=176) | Placebo (N=169)
Idiopathic thromnocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Anaesthetic complications (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCH 697243 (N=176) | Placebo (N=169)
Ear pruritus (Ear and labyrinth disorders) | 21 (35) | 1 (1)
Eye pruritis (Eye disorders) | 16 (17) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 5 (6) | 10 (19)
Lip swelling (Gastrointestinal disorders) | 13 (19) | 0 (0)
Oedema mouth (Gastrointestinal disorders) | 19 (29) | 1 (1)
Oral pruritis (Gastrointestinal disorders) | 68 (134) | 6 (11)
Stomatitis (Gastrointestinal disorders) | 26 (35) | 2 (2)
Pyrexia (General disorders) | 11 (12) | 12 (13)
Gastroenteritis viral (Infections and infestations) | 9 (10) | 6 (6)
Influenza (Infections and infestations) | 6 (6) | 10 (11)
Nasopharyngitis (Infections and infestations) | 33 (42) | 40 (58)
Sinusitis (Infections and infestations) | 6 (7) | 9 (9)
Upper respiratory tract infection (Infections and infestations) | 28 (42) | 26 (32)
Viral upper respiratory tract infection (Infections and infestations) | 14 (18) | 14 (18)
Headache (Nervous system disorders) | 23 (40) | 23 (38)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (20) | 19 (23)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (11) | 9 (12)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 13 (21) | 9 (12)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 27 (34) | 21 (27)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 13 (18) | 3 (5)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 9 (15) | 3 (4)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 65 (123) | 5 (9)
Uticaria (Skin and subcutaneous tissue disorders) | 9 (9) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results

of the study without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of publications that report any results of the study. The sponsor shall have the right to review and comment with respect to proprietary information, data accuracy, and fair balance in compliance with FDA regulations.